CLINICAL TRIAL: NCT01585961
Title: NAVISTAR® THERMOCOOL® SF Catheter: Observational Study in a Younger and Older Drug Refractory, Recurrent, Symptomatic Paroxysmal AF Population
Brief Title: NAVISTAR® THERMOCOOL® SF Catheter: Observational Study
Acronym: SFAF
Status: Completed | Type: Observational
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ThermoCool SF Phase IV
Record Dates: First submitted 2012-03-14; First posted 2012-04-26 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Atrial Fibrillation; Paroxysmal Arrhythmia
Keywords: Symptomatic paroxysmal; Atrial fibrillation; Observational; Acute procedural outcomes; Ablation; Drug refractory; Arrhythmia Recurrent; Symptomatic
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Catheter Ablation: These patients have drug refractory, recurrent, symptomatic paroxysmal atrial fibrillation, are aged 18 years or older, and have provided written informed consent to participate in the study, including consent to undergo catheter ablation with the study device.
  Interventions: Device: Catheter Ablation (NAVISTAR® THERMOCOOL® SF Catheter)

INTERVENTIONS:
Device: Catheter Ablation (NAVISTAR® THERMOCOOL® SF Catheter) — Administer anesthesia according to standard EP lab protocol, assess the fluid status of the subject (after each liter of infusate), determine if diuresis is necessary, and treat accordingly.

SUMMARY:
This is a prospective, interventional, observational, unblinded, single-arm, multicenter registry of younger and older subjects with drug refractory, recurrent, symptomatic paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
This study is to measure the "real-world" acute procedural outcomes (procedural efficiency, acute safety, and effectiveness at one year) associated with use of the NAVISTAR® THERMOCOOL® SF Catheter in a clinical setting in subjects with drug refractory, recurrent symptomatic paroxysmal atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Drug refractory, recurrent, symptomatic paroxysmal atrial fibrillation
* Age 18 years or older
* Patients must be able and willing to provide written informed consent to participate in the study

Exclusion Criteria:

* Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
* Previous ablation for atrial fibrillation
* Episodes of atrial fibrillation that last longer than 30 days and are terminated via cardioversion
* Uncontrolled heart failure, or NYHA Class III or IV heart failure
* Documented intra-atrial thrombus or other abnormality on pre-ablation echocardiogram
* Contraindication to anticoagulation
* Stroke, cardiac surgery, unstable angina, myocardial infarction or percutaneous coronary intervention within the past 3 months
* Awaiting cardiac transplantation
* Heart disease in which corrective surgery is anticipated within 6 months
* Enrollment in investigational drug, biologic or device study
* Subjects unwilling to comply with protocol or follow-up requirements
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Older and younger patients with drug refractory, symptomatic paroxysmal atrial fibrillation.
Sampling Method: Non-Probability Sample
Enrollment: 511 (Actual)
Dates: Start 2012-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gery Tomassoni, MD, Principal Investigator — Central Baptist Hospital; Scott Pollak, MD, Principal Investigator — Florida Hospital - Orlando; Andy Tran, MD, Principal Investigator — Scottsdale Healthcare Research Institute; Saumil Oza, MD, Principal Investigator — St. Vincent's Ambulatory Care, Inc.; Steven Compton, MD, Principal Investigator — Alaska Heart Institute, LLC; Anshul Patel, MD, Principal Investigator — St. Joseph's Hospital of Atlanta; Robert Fishel, MD, Principal Investigator — JFK Medical Center; Kenneth Civello, MD, Principal Investigator — Cardiovascular Research Foundation of Louisiana; Gaurang Gandhi, MD, Principal Investigator — Bethesda North Hospital; Alexandru Costea, MD, Principal Investigator — University of Cincinnati; Sreedhar Billakanty, MD, Principal Investigator — Riverside Methodist Hospital; H. James Wang, MD, Principal Investigator — Florida Hospital Memorial Medical Center; John Harding, MD, Principal Investigator — Central Bucks Specialists, Ltd.; Mohammed Khan, MD, Principal Investigator — Alexian Brothers Medical Center; Vijay Jayachandran, MD, Principal Investigator — Baylor All Saints Medical Center; Sree Karanam, MD, Principal Investigator — Lutheran Medical Group, LLC; M. Craig Delaughter, MD, Principal Investigator — Plaza Medical Center; Mohammad Jazayeri, MD, Principal Investigator — Bellin Memorial Hospital, Inc.; Abdi Rasekh, MD, Principal Investigator — Texas Heart Institute at St. Luke's Episcopal Hospital; Scott Allison, MD, Principal Investigator — Heart Center Research, LLC; Alexander Mazur, MD, Principal Investigator — University of Iowa Hospital & Clinics; Dhanunjaya Lakkireddy, MD, Principal Investigator — University of Kansas Hospitals; Alan Wimmer, MD, Principal Investigator — St. Luke's Hospital Mid American Heart Institute; Ali Hamzei, MD, Principal Investigator — Scripps Clinical Research; Shalin Shah, MD, Principal Investigator — Largo Medical Center; Michael Kutayli, MD, Principal Investigator — Bryan LGH Heart Institute; John Mandrola, MD, Principal Investigator — Baptist Hospital; Stuart Beldner, MD, Principal Investigator — North Shore University Hospital; Joshua Moss, MD, Principal Investigator — University of Chicago; Greg Bashian, MD, Principal Investigator — Centennial Heart; Patrick Whalen, MD, Principal Investigator — Vanderbilt Heart and Vascular Institute; Angelo Biviano, MD, Principal Investigator — New York Presbyterian Hospital, Columbia University Medical Center; Hussam Abuissa, MD, Principal Investigator — The Cardiac Center of Creighton University; Sumeet Mainigi, MD, Principal Investigator — Albert Einstein Medical Center; Charles Athill, MD, Principal Investigator — San Diego Cardiac Center; Edward Gerstenfeld, MD, Principal Investigator — UCSF Medical Center; Michael Chisner, MD, Principal Investigator — Cardiology Associates of Savannah; Vijendra Swarup, MD, Principal Investigator — Arizona Heart Hospital; Ziad Issa, MD, Principal Investigator — Prairie Education and Research Cooperative; Tariq Salam, MD, Principal Investigator — Cardiac Study Center; Sung Lee, MD, Principal Investigator — Washington Adventist Hospital; M. Magdy Migeed, MD, Principal Investigator — Genesis Healthcare Systems; Jonathan Sussman, MD, Principal Investigator — Morristown Medical Center; Bengt Herweg, MD, Principal Investigator — Tampa General Hospital; Pierce Vatterott, MD, Principal Investigator — United Heart and Vascular Clinic
Locations (45):
- United States (45):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Alaska Heart Institute, LLC, Anchorage, Alaska
  - Arizona Heart Hospital, Phoenix, Arizona
  - Scottsdale Healthcare Research Institute, Scottsdale, Arizona
  - Scripps Clinical Research, La Jolla, California
  - San Diego Cardiac Center, San Diego, California
  - UCSF Medical Center, San Francisco, California
  - JFK Medical Center, Atlantis, Florida
  - Florida Hospital Memorial Medical Center, Daytona Beach, Florida
  - St. Vincent's Ambulatory Care, Inc., Jacksonville, Florida
  - Largo Medical Center, Largo, Florida
  - Florida Hospital - Orlando, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - St. Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Cardiology Associates of Savannah, Savannah, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Lutheran Medical Group, LLC, Fort Wayne, Indiana
  - University of Iowa Hospital & Clinics, Iowa City, Iowa
  - University of Kansas Hospitals, Kansas City, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Baptist Hospital, Louisville, Kentucky
  - Cardiovascular Research Foundation of Louisiana, Baton Rouge, Louisiana
  - Washington Adventist Hospital, Takoma Park, Maryland
  - United Heart and Vascular Clinic, Saint Paul, Minnesota
  - St. Luke's Mid American Heart Institute, Kansas City, Missouri
  - Bryan LGH Heart Institute, Lincoln, Nebraska
  - The Cardiac Center of Creighton University, Omaha, Nebraska
  - Morristown Medical Center, Morristown, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - New York Presbyterian Hospital, Columbia University Medical Center, New York, New York
  - Bethesda North Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Genesis Healthcare Systems, Zanesville, Ohio
  - Central Bucks Specialists, LTD, Doylestown, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Centennial Heart, Nashville, Tennessee
  - Vanderbilt Heart and Vascular Institute, Nashville, Tennessee
  - Baylor All Saints Medical Center, Fort Worth, Texas
  - Plaza Medical Center, Grapevine, Texas
  - Texas Heart Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - Cardiac Study Center, Tacoma, Washington
  - Bellin Memorial Hospital, Inc., Green Bay, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Catheter Ablation: These patients have drug refractory, recurrent, symptomatic paroxysmal atrial fibrillation, are aged 18 years or older, and are able and willing to provide written informed consent to participate in the study.
  Catheter Ablation (NAVISTAR® THERMOCOOL® SF Catheter): Administer anesthesia according to standard EP lab protocol, assess the fluid status of the subject (after each liter of infusate), determine if diuresis is necessary, and treat accordingly.
Period: Overall Study
Arm/Group | Catheter Ablation
Started | 511
Safety | 508 (Patients ablated with study catheter)
Completed | 478
Not Completed | 33
Not completed — Death | 6
Not completed — Physician Decision | 1
Not completed — Decision to use non-study catheter | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 23
Not completed — Ablation cancelled for slow-heal wound | 1

BASELINE CHARACTERISTICS:
Population: Enrolled patients
Arm/Group | Catheter Ablation
Number analyzed (Participants) | 511
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 265
  >=65 years | 246
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194
  Male | 317
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 494
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 18
  White | 477
  More than one race | 2
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 511

OUTCOME MEASURES:

1. Primary Outcome: Total Fluoroscopy Time
Description: The fluoroscopy time will be measured for each phase (access, mapping, ablation, and validation) of the procedure and summed to derive the total time.
Time Frame: Day 0 (procedure)
Population: Subset of Safety Population with non-missing endpoint data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Catheter Ablation
Number analyzed (Participants) | 506
minutes | 26.4 (21.4)

2. Primary Outcome: Total Procedure Time
Time Frame: Day 0 (procedure)
Population: Subset of Safety Population with non-missing endpoint data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Catheter Ablation
Number analyzed (Participants) | 507
minutes | 169.8 (82.9)

3. Primary Outcome: Acute Procedural Success
Description: Confirmation of entrance and/or exit block across all targeted pulmonary veins.
Time Frame: Day 0 (procedure)
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Catheter Ablation
Number analyzed (Participants) | 508
participants | 488

4. Secondary Outcome: Mean Number of Radiofrequency (RF) Applications
Description: RF applications is defined as the number of times RF energy is delivered during the procedure.
Time Frame: Day 0 (procedure)
Population: Subset of Safety Population with non-missing endpoint data.
Measure: Mean (Standard Deviation); unit: number of applications
Arm/Group | Catheter Ablation
Number analyzed (Participants) | 489
number of applications | 45.0 (35.1)

5. Secondary Outcome: Total Radiofrequency (RF) Time
Description: Total RF time is defined as the total time that RF energy is delivered during the procedure.
Time Frame: Day 0 (procedure)
Population: Subset of Safety Population with non-missing endpoint data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Catheter Ablation
Number analyzed (Participants) | 505
minutes | 57.9 (37.0)

6. Secondary Outcome: Fluid Volume Delivered Via Ablation Catheter
Time Frame: Day 0 (procedure)
Population: Subset of Safety Population with non-missing endpoint data.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Catheter Ablation
Number analyzed (Participants) | 495
mL | 974.2 (481.8)

7. Secondary Outcome: Number of Patients With Repeat Ablations
Time Frame: 1 year
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Catheter Ablation
Number analyzed (Participants) | 508
participants | 74

8. Secondary Outcome: Post-procedure AF Symptoms
Description: Symptoms attributed to paroxysmal atrial fibrillation reported at 12 month visit
Time Frame: 12 Month Visit
Population: Subset of Safety Population with non-missing endpoint data.
Measure: Number; unit: participants
Arm/Group | Catheter Ablation
Number analyzed (Participants) | 470
participants | 155

9. Secondary Outcome: Number of Subjects With Lost Work Days, Related to AF, at 12 Month Visit
Time Frame: 12 Month Visit
Population: Subset of Safety Population with non-missing endpoint data.
Measure: Number; unit: participants
Arm/Group | Catheter Ablation
Number analyzed (Participants) | 477
participants | 20

10. Secondary Outcome: Number of Patients With Inpatient Hospital Visit(s) Related to Atrial Fibrillation
Time Frame: 12 Month Visit
Population: Population with Utilization Data
Measure: Number; unit: participants
Arm/Group | Catheter Ablation
Number analyzed (Participants) | 489
participants | 73

11. Secondary Outcome: Number of Patients With Outpatient Emergency Visits Related to Atrial Fibrillation
Time Frame: 12 Month Visit
Population: Population with Utilization Data
Measure: Number; unit: participants
Arm/Group | Catheter Ablation
Number analyzed (Participants) | 489
participants | 56

12. Secondary Outcome: Change in Atrial Fibrillation Effect on Quality of Life (AFEQT) Total Score
Description: Change is calculated as 12 month overall AFEQT score minus score at screening. An overall AFEQT score ranges from 0 to 100. A score of 0 corresponds to complete disability (or responding "extremely" limited, difficult or bothersome to all questions answered), while a score of 100 corresponds to no disability (or responding "not at all" limited, difficult or bothersome to all questions answered). Therefore a positive change in score corresponds to improvement in AF symptoms.
Time Frame: Screening to 12 Month Visit
Population: Subset of Safety Population with non-missing AFEQT data at 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Catheter Ablation
Number analyzed (Participants) | 462
units on a scale | 36.0 (23.7)

ADVERSE EVENTS:
Time Frame: Procedure through 7 days post-procedure
Arm/Group | Catheter Ablation
Serious Adverse Events (participants affected / at risk) | 63/508
Other Adverse Events (participants affected / at risk) | 79/508
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheter Ablation (N=508)
Atrial fibrillation (Cardiac disorders) | 9 (9)
Cardiac tamponade (Cardiac disorders) | 4 (4)
Pericardial effusion (Cardiac disorders) | 4 (4)
Pericarditis (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 3 (3)
Atrial tachycardia (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac perforation (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Catheter site hematoma (General disorders) | 3 (3)
Device difficult to use (foley) (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Subdural hematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
International normalized ratio decreased (Investigations) | 3 (3)
Electrocardiogram ST segment depression (Investigations) | 1 (1)
Hematocrit decreased (Investigations) | 1 (1)
Hemoglobin decreased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Syncope (Nervous system disorders) | 1 (1)
Transient global amnesia (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Femoral artery aneurysm (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Intra-abdominal hematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheter Ablation (N=508)
Atrial fibrillation (Cardiac disorders) | 15 (15)
Pericarditis (Cardiac disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 8 (8)
Pyrexia (General disorders) | 6 (6)
Catheter site hematoma (Injury, poisoning and procedural complications) | 11 (11)
Catheter site hemorrhage (Injury, poisoning and procedural complications) | 17 (17)
Fluid Overload (Metabolism and nutrition disorders) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11)
Dizziness (Nervous system disorders) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Hypotension (Vascular disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the Principal Investigator (PI)/Institution and the Sponsor (or its agents) that restricts the PI's rights to discuss, present, or publish trial results after the trial is completed. Please contact Biosense Webster for additional information.